CLINICAL TRIAL: NCT04349735
Title: Comparison of Three Methods of Assessment of INhalation TECHnique in Patients With Asthma and COPD
Brief Title: Comparison of 3 Methods to Assess Inhalation Technique
Acronym: CINTECH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Principal Investigator, Marta Dąbrowska, Principal Investigator, Medical University of Warsaw
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Inhalation technique 2
Record Dates: First submitted 2019-12-16; First posted 2020-04-16 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Asthma; COPD
Keywords: inhalation technique
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: comparison of three methods of assessment of inhaltion technique
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adults with asthma or COPD (Experimental): Assessment of inhalation technique by three methods in all patients
  Interventions: Other: Assessment of inhalation technique

INTERVENTIONS:
Other: Assessment of inhalation technique — Assessment of inhalation technique by 3 methods in every patient

SUMMARY:
A significant percentage of patients with asthma and COPD do not use their inhalers properly. Experts recommend that in patients with obstructive lung diseases, inhalation technique and patient adherence should be evaluated at every visit. The assessment of inhalation skills depends on the method of evaluation. There are few different methods of assessment of inhalation technique, however none of them is recommended as the most accurate.

Therefore, the aim of the study is:

1. to compare three different methods of assessment of inhalation technique in patients with asthma and COPD.

   These methods include:
   1. Checklist of mistakes in inhalation technique (including critical mistakes)
   2. 4 grade scale of inhalation technique
   3. Assessment by Vitalograph®AIM (Aerosol Inhaling Monitor)
2. to analyze the influence of Vitalograph®AIM based inhalation technique training on inhalation skills

One hundred and thirty patients with asthma or COPD, who use inhaled medication on a regular basis will be enrolled. Inhalation technique will be evaluated by two observers independently at the same time with all three methods (checklist, 4 grade scale, Vitalograph®AIM). To compare these methods, the investigators will analyze method reliability and validity. Additionally, inhalation technique will be evaluated 30 minutes after Vitalograph®AIM based training to analyze the potential benefit of its application in practicing inhalation skills.

DETAILED DESCRIPTION:
Asthma and chronic obstructive pulmonary disease (COPD) are common respiratory diseases. Inhaled therapy is the cornerstone of treatment in these two diseases. However, a significant proportion of patients with asthma and COPD do not use their inhalers properly. Experts recommend that in patients with obstructive lung diseases, inhalation technique and patient adherence should be evaluated at every visit, particularly before introducing changes to the patient's inhalation therapy. The assessment of inhalation skills depends on the method of evaluation. There are few different methods of assessment of inhalation technique, however, none of these methods is recommended as the most accurate.

Therefore, the aim of the study is:

1. to compare three different methods of assessment of inhalation technique in patients with asthma and COPD.

   These methods include:
   1. Checklist of mistakes in inhalation technique (including critical mistakes)
   2. 4 grade scale of inhalation technique
   3. Assessment by Vitalograph®AIM (Aerosol Inhaling Monitor)
2. to analyze an influence of using Vitalograph®AIM based inhalation technique training on inhalation skills.

Type of study: prospective, interventional, without randomization. Patients with asthma or COPD treated in hospital or in an out-patient clinic will be asked to participate in the study.

Study design One hundred and thirty patients with asthma or COPD, who use inhaled medication on a regular basis will be enrolled. Inhalation technique will be evaluated by two observers independently at the same time with all three methods (checklist, 4 grade scale, Vitalograph®AIM). To compare these methods, the investigators will analyze method reliability and validity. The reference assessment will be performed by two experienced pulmonologists.

Additionally, inhalation technique will be evaluated 30 minutes after Vitalograph®AIM based training to analyze the potential benefit of its application in practicing inhalation skills.

Outcomes

1. Comparison of three different methods of assessment of inhalation technique in patients with asthma and COPD (reliability, validity and accuracy)
2. Difference in the number of mistakes made during inhalation before and after the Vitalograph® AIM based training.

Investigators expect that results of this study will allow to identify the most accurate method for assessment of inhalation technique. Furthermore, the impact of Vitalograph®AIM based training on inhalation skills will be assessed..

ELIGIBILITY:
Inclusion criteria:

* informed consent for participating in the study
* age 18-85 years
* COPD or asthma diagnosed at least 3 months prior to enrollment
* using of at least one inhaler regularly every day
* using one of the inhalers: Metered Dose Inhalers (MDI), Dry Powder Inhalers (DPI) or Metered Dose Liquid Inhalers (MDLI)

Exclusion criteria:

* lack of informed consent
* age <18 years or > 85 years
* diagnosis of asthma or COPD not earlier than 3 months before enrollment
* using inhalers irregularly.
* symptoms of infection 5 days prior to beginning of the study
* comorbidity that could prevent patient from using Vitalograph®AIM to teach patient proper inhalation technique (i.e. advanced cognitive disorders, mental diseases, crucial neurological, vision or hearing disorders).

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2019-10-10 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Comparison of reliability of assessment of inhalation technique by checklist method in patients with asthma and COPD | baseline
  Assessment of reliability of checklist method measured by 2 observers by kappa Cohen coefficient
Comparison of reliability of assessment of inhalation technique by 4 grade scale in patients with asthma and COPD | baseline
  Assessment of reliability of 4 grade scale measured by 2 observers by kappa Cohen coefficient
Comparison of validity of assessment of inhalation technique by checklist method in patients with asthma and COPD | baseline
  Assessment of validity of checklist method measured by convergence between observer and an expert baseline by kappa Cohen coefficient
Comparison of validity of assessment of inhalation technique by 4 grade scale in patients with asthma and COPD | baseline
  Assessment of validity of 4 grade scale measured by convergence between observer and an expert baseline by kappa Cohen coefficient
Comparison of validity of assessment of inhalation technique by Vitalograph®AIM in patients with asthma and COPD | 30 minutes from baseline
  Assessment of validity of Vitalograph®AIM method (convergence between assessment of Vitalograph®AIM and an expert)

SECONDARY OUTCOMES:
Utility of Vitalograph® AIM in inhalation technique training | baseline and in 30 minutes
  Difference in number of inhalation mistakes before and after Vitalograph® AIM based training
Comparison of repeatability of assessment of inhalation technique by checklist method in patients with asthma and COPD | baseline and in 30 minutes
  Assessment of reliability of checklist method measured by 1 observer baseline and in 30 minutes by kappa Cohen coefficient
Comparison of repeatability of assessment of inhalation technique by 4 grade scale in patients with asthma and COPD | baseline and in 30 minutes
  Assessment of reliability of 4 grade scale measured by 1 observer baseline and in 30 minutes by kappa Cohen coefficient

CONTACTS AND LOCATIONS:
Overall Officials: Rafał Krenke, MD,PhD,Prof, Study Director — Medical University of Warsaw
Locations (1):
- Department of Internal Medicine, Pneumonology and Allergology, Medical University of Warsaw, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Usmani OS, Lavorini F, Marshall J, Dunlop WCN, Heron L, Farrington E, Dekhuijzen R. Critical inhaler errors in asthma and COPD: a systematic review of impact on health outcomes. Respir Res. 2018 Jan 16;19(1):10. doi: 10.1186/s12931-017-0710-y. PMID 29338792
- [Result] Laube BL, Janssens HM, de Jongh FH, Devadason SG, Dhand R, Diot P, Everard ML, Horvath I, Navalesi P, Voshaar T, Chrystyn H; European Respiratory Society; International Society for Aerosols in Medicine. What the pulmonary specialist should know about the new inhalation therapies. Eur Respir J. 2011 Jun;37(6):1308-31. doi: 10.1183/09031936.00166410. Epub 2011 Feb 10. PMID 21310878
- [Result] Melani AS, Bonavia M, Cilenti V, Cinti C, Lodi M, Martucci P, Serra M, Scichilone N, Sestini P, Aliani M, Neri M; Gruppo Educazionale Associazione Italiana Pneumologi Ospedalieri. Inhaler mishandling remains common in real life and is associated with reduced disease control. Respir Med. 2011 Jun;105(6):930-8. doi: 10.1016/j.rmed.2011.01.005. Epub 2011 Mar 2. PMID 21367593
- [Result] Sanchis J, Gich I, Pedersen S; Aerosol Drug Management Improvement Team (ADMIT). Systematic Review of Errors in Inhaler Use: Has Patient Technique Improved Over Time? Chest. 2016 Aug;150(2):394-406. doi: 10.1016/j.chest.2016.03.041. Epub 2016 Apr 7. PMID 27060726